CLINICAL TRIAL: NCT04313985
Title: Electrical Stimulation as an Adjunctive Therapy to Increase Vascular Perfusion in People With PAD or PVD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI relocated
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 45628
Record Dates: First submitted 2019-08-01; First posted 2020-03-18 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: PAD - Peripheral Arterial Disease; PVD- Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both the participant and the care provider will be masked as to what treatment the participant is receiving during each study visit. Only the study coordinator will know which treatment is being conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electrical Stimulation First, then Sham Stimulation (Active Comparator): Treat the patient's wound area:
  Place self-adhesive, conductive electrode pads on either side of the wound on the skin where the pads are not placed in the open wound itself, but rather in the surrounding area with one pad on each side of the wound.
  Connect the pads to the lead wire to the Avazzia device. Turn on the Avazzia device and change modes to the RSI mode. Increase power to maximum comfortable power level for the patient. If the patient cannot feel the output, then increase power to 250.
  Instruct the patient to reduce the power level if it begins to feel too strong. (sometimes as the microstimulation is applied, the tissue will become more sensitive to the stimulation. In this case the power should be reduced for patient comfort.) Allow to run unattended for 15 minutes. Take a picture of the pad placement and display on the device to document location, power setting, and treatment mode while the treatment is running for the 15 minutes.
  Interventions: Device: Tennant Biomodulator-Pro™ Device
- Sham Electrical Stimulation First, then Electrical Stimulation (Sham Comparator): Treat the patient's wound area:
  Place self-adhesive, conductive electrode pads on either side of the wound on the skin where the pads are not placed in the open wound itself, but rather in the surrounding area with one pad on each side of the wound.
  Connect the pads to the lead wire to the Avazzia device. Turn on the Avazzia device and change modes to the RSI mode. Increase power to maximum comfortable power level for the patient. If the patient cannot feel the output, then increase power to 250.
  Instruct the patient to reduce the power level if it begins to feel too strong. (sometimes as the microstimulation is applied, the tissue will become more sensitive to the stimulation. In this case the power should be reduced for patient comfort.) Allow to run unattended for 15 minutes. Take a picture of the pad placement and display on the device to document location, power setting, and treatment mode while the treatment is running for the 15 minutes.
  Interventions: Device: Tennant Biomodulator-Pro™ Device

INTERVENTIONS:
Device: Tennant Biomodulator-Pro™ Device — Tennant Biomodulator-Pro™ conductive electrode pads will be placed on both sides of the wound. The device will either deliver electrical stimulation or no stimulation depending on treatment period.

SUMMARY:
The purpose of this study is to apply Avazzia micro-current stimulation to patients with chronic, non-healing wounds to determine if this therapy is effective in perfusion and bacterial measurements.

DETAILED DESCRIPTION:
Investigators hope to learn if micro-current stimulation to a chronic, non-healing wound can be lead to healing. Perfusion studies and bacterial measurements will be assessed before and after treatment on this cross-over study.

Avazzia microcurrent stimulation was applied to patients with chronic, non-healing wounds in Malaysia and was presented at the international wound conference. In 2015 a poster presentation was presented with a 10-patient case series, and in August 2016, a presentation was made by Dr. Nair, keynote speaker about his 100- patient case series showing that the treatment was safe and effective. Dr. Nair followed this study with a 5-patient study looking at perfusion images using SPY- LUNA imaging equipment. The 5-patient study looked at different methods of applying the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a chronic non-healing wound that has not healed in 30 days in their feet, legs, lower back or buttocks, but not in their hands because the hands will be used to verify equipment operation.
* Age ≥18 and ≤70 years
* Wound area is ≥0.5 cm2 and ≤22 cm2
* Willing and able to comply with weekly visits to clinic (e.g., reliable transportation)

Exclusion Criteria:

* Presence of an electrical implant such as a cardiac pacemaker or neural stimulator
* Patient is currently pregnant, possibly pregnant or breast-feeding User of any microcurrent device in the past six (6) months prior to enrollment in the study
* Patient is experiencing a medical emergency
* Patient is diagnosed with neuropathy from sources other than diabetes, such as heavy metal, xenobiotic toxicity
* Patient is diagnosed with Charcot-Marie-Tooth or similar genetically inheritable neuropathic disease(s)
* Patient is diagnosed with end-stage kidney disease/dialysis or severe kidney insufficiency
* Patient is diagnosed with malignancies (cancers) undergoing treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C Gurtner, MD, Principal Investigator — Stanford University School of Medicine- Plastic & Reconstructive Surgery
Locations (1):
- Stanford Advanced Wound Care Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrical Stimulation First, Then Sham Stimulation; Sham Stimulation First, the Electrical Stimulation: Tennant Biomodulator-Pro™ conductive electrode pads placed on both sides of the wound, delivering electrical stimulation or no stimulation in the respective study period.
Period: Treatment Period 1 (1 Week)
Arm/Group | Electrical Stimulation First, Then Sham Stimulation | Sham Stimulation First, the Electrical Stimulation
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Treatment Period 2 (1 Week)
Arm/Group | Electrical Stimulation First, Then Sham Stimulation | Sham Stimulation First, the Electrical Stimulation
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Follow-up Period (1 Week)
Arm/Group | Electrical Stimulation First, Then Sham Stimulation | Sham Stimulation First, the Electrical Stimulation
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electrical Stimulation First, Then Sham Stimulation | Sham Stimulation First, the Electrical Stimulation | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4
Pain Score [Mean (Standard Deviation); unit: score on a scale] — Measured on a numerical 0-10 visual scale (0 = no pain, 10 = worst pain imaginable)
  score on a scale | 0 (0) | 2.5 (3.536) | 1.25 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Wound Tissue Perfusion
Description: To compare wound tissue perfusion following treatment vs placebo (as measured using the HyperMed HyperView device)
Time Frame: Day 7 of the respective treatment period
Population: Data were not collected for the outcome measure.
Groups:
- Electrical Stimulation: Tennant Biomodulator-Pro™ conductive electrode pads placed on both sides of the wound delivering electrical stimulation.
- Sham Electrical Stimulation: Tennant Biomodulator-Pro™ conductive electrode pads placed on both sides of the wound delivering no stimulation.
Arm/Group | Electrical Stimulation | Sham Electrical Stimulation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Change in Wound Area as a Measure of Healing Rate
Description: To compare rate of wound healing following treatment vs placebo (measured as percentage change in wound area).
Time Frame: Day 7 of the respective treatment period
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Electrical Stimulation | Sham Electrical Stimulation
Number analyzed (Participants) | 4 | 4
percentage change | -31 [-71 to 19] | -52 [-65 to 38]

3. Secondary Outcome: Bacterial Biopsies
Description: To compare bacterial burden at the wound site following treatment vs placebo (measured in cells per gram of wound tissue from quantitative deep tissue swab)
Time Frame: From time of randomization up until wound healing or 3 weeks, whichever came first
Population: Data were not collected for this outcome measure.
Arm/Group | Electrical Stimulation | Sham Electrical Stimulation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pain Score
Description: To compare patient pain at the wound site following treatment vs placebo, measured on a numerical 0-10 visual scale (0 = no pain, 10 = worst pain imaginable)
Time Frame: Day 7 of the respective treatment period
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Electrical Stimulation | Sham Electrical Stimulation
Number analyzed (Participants) | 4 | 4
score on a scale | 0 [0 to 1.75] | 1 [0 to 1.25]

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Electrical Stimulation | Sham Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
This study fell far short of it's planned enrollment size and failed to achieve statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT04313985/Prot_SAP_000.pdf